CLINICAL TRIAL: NCT05212792
Title: Genomics of COVID-19 Vaccine-induced Adverse Events (Guillain-Barré Syndrome [GBS], Vaccine-induced Immune Thrombotic Thrombocytopenia [VITT]/thrombosis with Thrombocytopenia Syndrome [TTS], and Myocarditis/pericarditis)
Brief Title: Genomics and COVID-19 Vaccine Adverse Events
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bruce Carleton, Director, Pharmaceutical Outcomes Programme, BC Children's Hospital; Division Head, Translational Therapeutics, Department of Pediatrics, University of British Columbia, University of British Columbia
Other Study IDs: H21-03404
Record Dates: First submitted 2022-01-25; First posted 2022-01-28 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Vaccine Adverse Reaction
Keywords: Genomics; COVID-19 vaccine adverse event; Guillain-Barré syndrome (GBS); Vaccine-induced Immune Thrombotic Thrombocytopenia (VITT); Thrombosis with thrombocytopenia syndrome (TTS); Myocarditis; Pericarditis
MeSH Terms: conditions — Guillain-Barre Syndrome; Myocarditis; Pericarditis | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Case with COVID-19 vaccine adverse event: Patients with GBS, VITT/TTS, or myocarditis/pericarditis after COVID-19 vaccination
  Interventions: Biological: COVID-19 vaccines
- Control without COVID-19 vaccine adverse event: Participants without experiencing GBS, VITT/TTS, or myocarditis/pericarditis after COVID-19 vaccination
  Interventions: Biological: COVID-19 vaccines

INTERVENTIONS:
Biological: COVID-19 vaccines — Any licensing COVID-19 vaccine platform

SUMMARY:
Vaccines routinely used are extremely safe; however, severe adverse events to vaccines do occur. As vaccination against COVID-19 has begun, adverse events to the vaccine, particularly Guillain-Barré syndrome (GBS), vaccine-induced immune thrombotic thrombocytopenia (VITT)/thrombosis with thrombocytopenia syndrome (TTS), and myocarditis/pericarditis, after COVID-19 vaccination have been reported worldwide.

Study hypothesis: there are genetic factors that contribute to increased risks of particular COVID-19 vaccine-induced adverse events.

The objective of the study is to determine if there are specific genetic factors strongly associated with each of the COVID-19 vaccine-induced adverse events (i.e., GBS, VITT/TTS, and myocarditis/pericarditis).

DETAILED DESCRIPTION:
Purpose:

Reduce the risk of COVID-19 vaccine-induced adverse events (i.e., GBS, VITT/TTS, and myocarditis/pericarditis) through improved understanding of the biology underlying these severe adverse events and the genetic contribution to their cause

Research Design:

* Prospective case-control study designs will be performed to investigate the genetic associations of Guillain-Barré syndrome (GBS), vaccine-induced immune thrombotic thrombocytopenia (VITT)/thrombosis with thrombocytopenia syndrome (TTS), and myocarditis/pericarditis strongly associated (OR ≥ 3.0) with COVID-19 vaccination.
* Determined cases of specific COVID-19 vaccine-induced GBS, VITT/TTS, and myocarditis/pericarditis, and vaccinated controls without these adverse events will be included.
* Saliva DNA samples from eligible adverse event cases and vaccinated controls will be collected.
* Candidate gene and genome-wide association studies (GWAS) approaches will be conducted.
* Genomics analyses will be stratified by severity, age, sex, vaccine, and other critical covariates as determined by the GVDN Work Group for each adverse event and as adequately powered analyses allow.
* To complement GWAS, particularly in protein-coding regions, additional whole-exome sequencing (WES) will be performed on the most severe patients who are categorized as Brighton Collaboration Level One case of COVID-19 vaccine-induced adverse events to identify the most possible disease-causing mutations.

ELIGIBILITY:
Inclusion Criteria:

* Case: Any patient who received COVID-19 vaccines and developed GBS, VITT/TTS, or myocarditis/pericarditis after vaccination
* Control: Any participant who received COVID-19 vaccines and does not experience GBS, VITT/TTS, or myocarditis/pericarditis.

Exclusion Criteria:

* Individuals who have not received a COVID-19 vaccine
* Individuals who are unable to provide informed consent

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any individual who received a COVID-19 vaccine.
  A total of 825 adverse event cases (n=275 each for GBS, VITT/TTS, and myocarditis/pericarditis) and 5,500 vaccine-matched controls (n=2,750 each for mRNA and adenovirus vector COVID-19 vaccine platforms) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 6325 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Determine specific genetic factors associated with particular COVID-19 vaccine-induced Guillain-Barré syndrome (GBS), vaccine-induced immune thrombotic thrombocytopenia (VITT)/thrombosis with thrombocytopenia syndrome (TTS), and myocarditis/pericarditis | December 2025

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Carleton, PharmD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- See also: Global Vaccine Data Network and project information — https://www.globalvaccinedatanetwork.org/